CLINICAL TRIAL: NCT07162428
Title: The Effect of Art Therapy on Disease Severity and Anxiety Levels in Inpatients at a Psychiatry Clinic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: tugbasahin
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the art therapy intervention group or the control group receiving standard care
Masking Description: This is an open-label study; neither participants nor investigators are blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Art Therapy Intervention (Experimental): Participants in this group will receive art therapy sessions in addition to standard psychiatric care. The intervention will consist of 3 sessions per week, conducted on 5 consecutive days, with each session lasting approximately 50 minutes. Sessions will be carried out in groups of 8 participants and will focus on creative expression through drawing and painting. All sessions will be facilitated by a trained art therapist.
  Interventions: Behavioral: Art Therapy
- Control Group (Standard Care) (No Intervention): Participants in this group will receive standard psychiatric care without additional art therapy sessions.

INTERVENTIONS:
Behavioral: Art Therapy — The art therapy sessions will be conducted by a certified art therapist who has completed a two-year training program, together with a psychiatric nurse who has completed a 4-hour training course on "Severe Personality Disorders and Therapeutic Interventions - Art Therapy." A clinical nurse and a psychiatry resident will also participate as observers. The therapist will deliver the intervention through semi-structured sessions, following a predefined content and method. These sessions are referred to as Semi-Structured Art Therapy Sessions.
  Arms: Art Therapy Intervention

SUMMARY:
The aim of this study is to examine the effect of art therapy applied to inpatients in the psychiatry ward on disease severity and anxiety levels. Art therapy is considered a complementary intervention that can positively contribute to the psychiatric recovery process by facilitating the expression and regulation of an individual's emotional state.

This research will be conducted with a randomized controlled design and aims to demonstrate the effectiveness of art therapy practices within the clinical process through objective data. The originality of the study lies in the fact that art therapy will be implemented with individuals hospitalized in an acute psychiatric ward. In this respect, the study provides the opportunity to evaluate the applicability of art therapy even during crisis periods and carries the potential to make significant practice-oriented contributions to the field of mental health.

DETAILED DESCRIPTION:
Mental health is currently defined as a significant public health issue on a global scale. Mental disorders manifest across a wide spectrum, ranging from mild anxiety disorders to behavioral abnormalities. Psychiatric illnesses not only diminish individuals' quality of life but also impose substantial social and economic burdens on healthcare systems.

Alternative and complementary treatment methods are gaining increasing importance in alleviating this burden. In this context, art therapy has recently attracted attention as a supportive method in psychiatric treatments. The British Association of Art Therapists (BAAT) defines art therapy as "a form of psychotherapy in which art materials are used as the primary medium of expression and communication," whereas the American Art Therapy Association (AATA) defines it as "a mental health and human services profession that integrates creative processes, psychological theory, and human experience".

Art therapy represents a multidimensional approach that encompasses various practices such as drama therapy, dance-movement psychotherapy, body therapy, music therapy, painting, drawing, and crafts. This form of therapy aims to promote recovery not only at the mental level but also at the physical and emotional levels in the treatment of psychiatric disorders .

Research has shown that art therapy enhances individual expressive abilities, facilitates emotion regulation, and provides a personalized healing process. It has been demonstrated to yield effective results particularly in post-traumatic stress disorder (PTSD), personality disorders, and mood disorders. Furthermore, its effectiveness in reducing depression in elderly individuals has been supported by randomized controlled trials. Similarly, studies on reducing anxiety levels in children have also reported positive outcomes.

This study aims to investigate the effect of art therapy practices on disease severity and anxiety levels among inpatients in a psychiatric ward, using a randomized controlled trial design. The originality of this study lies in its implementation of art therapy with individuals hospitalized in an acute psychiatric ward. In this regard, examining the direct impact of art therapy within the clinical process has the potential to provide significant practical contributions for both practitioners and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older.

Currently hospitalized in the psychiatry clinic and expected to remain hospitalized during the study period.

No medical condition such as intellectual disability or organic mental disorder that would interfere with the administration of scales and tests.

A PANSS score of ≤62 (since a score of 61 is considered the remission criterion in schizophrenia, patients scoring 62 or below will be included).

A score between 5-18 on the Young Mania Rating Scale.

Receiving treatment in the clinic for at least 3 days.

Providing verbal and/or written informed consent to participate in the study.

Exclusion Criteria:

Being in an acute psychotic episode or having severe psychotic symptoms (e.g., severe delusions, hallucinations) making the patient unsuitable for group participation.

Clinical conditions involving excessive agitation or homicidal risk that make group participation inappropriate.

Inability to actively participate in art therapy due to visual, hearing, or severe motor impairments.

Patients for whom discharge is planned during the clinical course (e.g., those scheduled for discharge in less than 3 days).

Diagnosis of an organic mental disorder (e.g., dementia, delirium).

Severe physical illness or motor impairment preventing participation in group activities

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-09-16 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS) | Before and after each therapy session (daily assessments during the 5-day intervention week for each group). Each group receives one week of therapy; in total, three groups will complete the intervention over three consecutive weeks.
  The YMRS is an 11-item scale developed by Young et al. to assess the severity of manic episodes. Seven items are rated on a 5-point Likert scale and four items on a 9-point Likert scale, with a total score range of 0 to 44. The Turkish version has been validated for reliability and validity. The total score can range from 0 to 60, with higher scores indicating more severe manic symptoms.
State-Trait Anxiety Inventory (STAI - Form I and II) | Before and after each session across the 5-day intervention week for each group (three groups in total, over three weeks).
  Self-report measure assessing state and trait anxiety, consisting of 20 items each, rated on a 4-point Likert scale.
Positive and Negative Syndrome Scale (PANSS) | Before and after each session across the 5-day intervention week for each group (three groups in total, over three weeks).
  The PANSS is a 30-item scale developed by Kay et al. to assess positive symptoms, negative symptoms, and general psychopathology in schizophrenia. Scores are rated across three subscales. The Turkish version has been validated by Kostakoğlu et al. In this scale (PANSS: Positive and Negative Syndrome Scale), as the score increases, symptoms/psychopathology become more severe. In other words, the higher the score, the greater the severity of symptoms and the greater the impairment in the patient's daily functioning.

IPD SHARING:
Plan to Share IPD: No